CLINICAL TRIAL: NCT01920919
Title: Low-dose Dexamethasone in Newly Diagnosed Pulmonary Sarcoidosis
Acronym: DEXSAR
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: St. Antonius Hospital (Other)
Responsible Party: Principal Investigator, R Vis, Hospital Pharmacist, St. Antonius Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2013-000242-18
Record Dates: First submitted 2013-08-07; First posted 2013-08-12 (Estimated); Last update posted 2014-11-19 (Estimated); Status verified 2014-11

CONDITIONS: Sarcoidosis
MeSH Terms: conditions — Sarcoidosis | interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Dexamethasone 1 mg (Experimental): Dexamethasone 1 mg per day, for 180 days
  Interventions: Drug: Dexamethasone
- Placebo (Placebo Comparator): Placebo tablet, for 180 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dexamethasone
  Arms: Dexamethasone 1 mg
Drug: Placebo
  Arms: Placebo

SUMMARY:
This trial examines whether low grade suppression of the initial inflammatory process of sarcoidosis by intervention with low-dose dexamethasone therapy achieves significant alleviation of (sub-)acute symptoms, improvement in quality of life, increase in work productivity, and whether this intervention prevents disease progression and reduces total health-care costs.

DETAILED DESCRIPTION:
The orphan disease sarcoidosis causes a major reduction in quality of life and loss of work productivity, especially in young adults. Most patients are diagnosed between the age of 20-40 years. In sarcoidosis, multiple organs are affected by inflammation; the cause of the disease is unknown and no curative medication exists. Sarcoidosis invalidates the lives of most patient for many years.

Although curative (pharmaco) therapy is not on hand, immunosuppressive drugs may control the symptoms of the disease. These symptoms are caused by the inflammation in multiple organs, foremost the lungs and the lymphoid system. However, 90% of the sarcoidosis patients receives no immunosuppressive medication at all during the first months after diagnosis, even though the immune system is then highly activated and patients suffer from severe complaints like malaise, fatigue and pain. This wait-and-see policy is common international practice, but scientific grounds and official guidelines are lacking.

This project examines whether low grade suppression of the initial inflammatory process of sarcoidosis by intervention with low-dose dexamethasone therapy achieves significant alleviation of (sub-)acute symptoms, improvement in quality of life, increase in work productivity, and whether this intervention prevents disease progression and reduces total health-care costs.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of sarcoidosis, confirmed by histology or cytology
* Age 18-60 years
* No affected organ requiring high dose immunosuppressive therapy
* Short Form - 36 subscale physical functioning score < 70 points

Exclusion Criteria:

* Allergy to corticosteroids
* Diagnosis of glaucoma, osteoporosis, history of fractures
* History of gastric ulcera in the past 12 months
* Current use of Non Steroidal Anti Inflammatory Drug without co-prescription of Proton Pump Inhibitor
* Current use of carbamazepin, fenytoin, rifampicin
* Obesity (BMI > 30)
* Pregnancy of lactation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 76 (Estimated)
Dates: Start 2013-06; Primary Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Change in health-related quality of life versus baseline | 0, 3, 6, 12, 18, 24 months
  The primary outcome measure is the change in health-related quality of life compared with baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- St Antonius Hospital, Nieuwegein, Netherlands